CLINICAL TRIAL: NCT01842295
Title: Bariatric Surgery, Nutrition, and Sperm Quality of Adult Obese Men on Childbearing Age : A Multicentric Cohort Study
Brief Title: Bariatric Surgery and Sperm Quality
Acronym: BARIASPERM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: P110153; AOM11193 (Other Grant/Funding Number: Programme Hospitalier de Recherche Clinique (PHRC))
Record Dates: First submitted 2013-02-19; First posted 2013-04-29 (Estimated); Last update posted 2025-09-11 (Actual); Status verified 2025-09

CONDITIONS: Obesity; Bariatric Surgery
Keywords: Obesity; Bariatric surgery; Sperm quality; Fertility
MeSH Terms: conditions — Obesity | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bariatric surgery (No Intervention): Obese men with associated co-morbidities selected for bariatric surgery by multidisciplinary team
  Interventions: Other: Blood and sperm samples

INTERVENTIONS:
Other: Blood and sperm samples — Blood and sperm samples will be done in each visit

SUMMARY:
The purpose of this study is to evaluate the impact of a bariatric surgery (gastric banding, bypass, sleeve gastrectomy) on several parameters (quality of sperm and others biological parameters, lifestyle, quality of life) involved in fertility of obese adult men.

DETAILED DESCRIPTION:
In order to assess how bariatric surgery may influence their fertility parameters, patients will attend to 3 visits :

First visit (inclusion, before surgery) :

* Signature of consent
* Patient interview (Collection of data on background, treatments, socio-demographic characteristics, social and familial environment, food consumption and habits, tobacco and alcohol use, physical activity, libido and quality of life (surveys))
* Clinical examination and anthropometric assessment (BMI, blood pressure, expired CO)
* Blood samples (Metabolic and nutritional plasmatic biomarkers ; Plasmatic oxidative stress biomarkers ; antioxidants micronutrients ; hormones of adiposity and inflammation ; sex hormones ; persistent contaminants)
* Sperm sample (sperm count-morphology ; DNA fragmentation ; CASA)

Bariatric surgery

Second visit (6 month follow-up)

* Report of adverse events if any
* Surveys
* Blood and sperm samples

Third visit (12 month follow-up)

* Report of adverse events if any
* Blood and sperm samples

ELIGIBILITY:
Inclusion Criteria:

* Obese men with BMI ≥ 40kg/m² or 35 kg/m² with associated co-morbidities
* Selected for bariatric surgery by multidisciplinary team
* From 18 to 50 years old included
* With a first medical consultation and its results
* With their written informed consent to participate in the study
* No problem for understanding verbal or written French
* An affiliation to social security

Exclusion Criteria:

* Not candidates for surgery
* With non idiopathic alteration of spermatogenesis

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2013-02-15 (Actual); Primary Completion 2016-03-25 (Actual); Study Completion 2016-03-25 (Actual)

PRIMARY OUTCOMES:
Number of total spermatozoids (NTS) variation | 6 months after surgery
  Comparison before/after surgery

SECONDARY OUTCOMES:
Number of total spermatozoids (NTS) variation | 1 year after surgery
  Comparison before/after surgery
sperm caracteristics | 6 months and 1 year after surgery
  Comparison before/after surgery
Effect of biological parameters on NTS variation | 6 months and 1 year after surgery
  Comparison before/after surgery and search of correlation
Evaluation of environmental parameters : physical activity | 6 months and 1 year after surgery
  Comparison before/after surgery
Other spermatic parameters : DNA fragmentation | 6 months and 1 year after surgery
  Comparison before/after surgery
Other spermatic parameters : CASA | 6 months and 1 year after surgery
  Comparison before/after surgery
Effect of anthropometric parameters on NTS variation | 6 months and 1 year after surgery
  Comparison before/after surgery and search of correlation
Evaluation of environmental parameters : tobacco consumption | 6 months and 1 year after surgery
  Comparison before/after surgery
Evaluation of environmental parameters : libido | 6 months and 1 year after surgery
  Comparison before/after surgery
Evaluation of environmental parameters : quality of life | 6 months and 1 year after surgery
  Comparison before/after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Levy, MD, Study Chair — Jean Verdier Hospital
Locations (1):
- Jean Verdier Hospital, Bondy, France

REFERENCES:
- [Background] Carette C, Levy R, Eustache F, Baron G, Coupaye M, Msika S, Barrat C, Cohen R, Catheline JM, Brugnon F, Slim K, Barsamian C, Chevallier JM, Bretault M, Bouillot JL, Antignac JP, Rives-Lange C, Ravaud P, Czernichow S. Changes in total sperm count after gastric bypass and sleeve gastrectomy: the BARIASPERM prospective study. Surg Obes Relat Dis. 2019 Aug;15(8):1271-1279. doi: 10.1016/j.soard.2019.04.019. Epub 2019 Apr 25. PMID 31147284
- [Background] Mifsud F, Czernichow S, Carette C, Levy R, Ravaud P, Cynober L, Neveux N, Rives-Lange C; Bariasperm Study Group. Behaviour of plasma citrulline after bariatric surgery in the BARIASPERM cohort. Clin Nutr. 2021 Feb;40(2):505-510. doi: 10.1016/j.clnu.2020.05.045. Epub 2020 Jun 12. PMID 32891457
- [Background] di Frega AS, Dale B, Di Matteo L, Wilding M. Secondary male factor infertility after Roux-en-Y gastric bypass for morbid obesity: case report. Hum Reprod. 2005 Apr;20(4):997-8. doi: 10.1093/humrep/deh707. Epub 2004 Dec 23. PMID 15618249
- [Background] MacDonald AA, Herbison GP, Showell M, Farquhar CM. The impact of body mass index on semen parameters and reproductive hormones in human males: a systematic review with meta-analysis. Hum Reprod Update. 2010 May-Jun;16(3):293-311. doi: 10.1093/humupd/dmp047. Epub 2009 Nov 4. PMID 19889752
- [Background] Sermondade N, Massin N, Boitrelle F, Pfeffer J, Eustache F, Sifer C, Czernichow S, Levy R. Sperm parameters and male fertility after bariatric surgery: three case series. Reprod Biomed Online. 2012 Feb;24(2):206-10. doi: 10.1016/j.rbmo.2011.10.014. Epub 2011 Nov 3. PMID 22196889